CLINICAL TRIAL: NCT01743040
Title: Pivotal Study of the CADence Device in Detection of Coronary Artery Diseases
Brief Title: Clinical Evaluation of the CADence Device in Detection of Coronary Artery Diseases
Acronym: TURBULENCE
Status: Completed | Type: Observational
Sponsor: AUM Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1038-001
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Nuclear Stress Test; CT Angiography; Angiography; CADence
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CADence plus Standard Angiogram: All patients who were indicated for angiogram due to results of SPECT nuclear stress test
  Interventions: Diagnostic Test: CADence
- CADence plus CT Angiogram: All patients who were not indicated for angiogram due to results of SPECT nuclear stress test underwent CT angiogram
  Interventions: Diagnostic Test: CADence

INTERVENTIONS:
Diagnostic Test: CADence — Patients with chest pain and two or more coronary risk factors and who were already indicated for nuclear stress test were enrolled in the study. The CADence was performed prior to nuclear stress test. Patients underwent standard angiogram based upon normal clinical judgement. In all other patients a CT angiogram followed.
  CADence is a handheld equipped with acoustic sensor technology, a patient booklet, remote algorithm and final report.
  Other Names: CT Angiogram; Angiogram; Nuclear Stress Test

SUMMARY:
This is a multi-center, prospective, non-randomized, double-blinded trial to evaluate the sensitivity and specificity of the CADence device in detecting the existence of clinically significant coronary artery disease as determined by either standard or CT angiography.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-randomized, double-blinded, trial to evaluate the performance of the CADence in detecting the existence of at least one major coronary artery with clinically significant stenosis in a subject is defined as the presence of at least one lesion with ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending, mid Left anterior Descending, proximal Left Circumflex, mid Left Circumflex , proximal Right Coronary Artery, mid Right Coronary Artery, distal Right Coronary Artery and Obtuse Margin 1, Obtuse Margin 2, and Ramus Intermedius if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left Main coronary arteries.

Consented subjects will be evaluated with the CADence device and then undergo nuclear stress testing followed by either computed tomography or standard coronary angiography. The maximum expected timeframe between CADence and computed tomography Angiography or standard angiography is 6 weeks.

This is a double-blinded study. All physicians and subjects will be masked to the diagnostic results of the CADence until completion of CADence, nuclear stress, computed tomography or standard coronary angiogram testing for the subjects. Patient care will not be based on the CADence results.

Study participation will conclude after the computed tomography angiography or standard coronary angiography procedure.

computed tomograph or standard coronary angiography are considered acceptable clinical reference standards in this study and are gold standards for detection of coronary artery disease. The experimental unit of this study is the subject. Existence of clinically significant coronary artery disease in a subject is defined as the presence of at least one lesion with ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending, mid Left anterior Descending, proximal Left Circumflex, mid Left Circumflex, proximal Right Coronary Artery, mid Right Coronary Artery, distal Right Coronary Artery and Obtuse Margin 1, Obtuse Margin 2, and Ramus Intermedius if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left Main coronary arteries.

The study required sample size is 826 but may enroll up to 1,300 subjects. The sensitivity and specificity of the CADence are expected to be 80% and 73% respectively. Observed sensitivity and specificity will be compared to nuclear stress literature-based performance standards of 83% and 80% respectively using one sample non-inferiority binomial tests with a non-inferiority margin of 15 percentage points. Sample size requirements are 109 subjects with the presence of at least one lesion with ≥ ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending, mid Left anterior Descending, proximal Left Circumflex, mid Left Circumflex, proximal Right Coronary Artery, mid Right Coronary Artery, distal Right Coronary Artery and Obtuse Margin 1, Obtuse Margin 2, and Ramus Intermedius if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left MAIN coronary arteries. to test the sensitivity hypothesis and 268 subjects without the presence of at least one lesion with ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending, mid Left anterior Descending, proximal Left Circumflex, mid Left Circumflex, proximal Right Coronary Artery, mid Right Coronary Artery, distal Right Coronary Artery and Obtuse Margin 1, Obtuse Margin 2, and Ramus Intermedius if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left MAIN coronary arteries. to test the specificity hypothesis. It was assumed that 15 percent of enrolled subjects would be found to have the presence of at least one lesion with ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending, mid Left anterior Descending, proximal Left Circumflex, mid Left Circumflex, proximal Right Coronary Artery, mid Right Coronary Artery, distal Right Coronary Artery and Obtuse Margin 1, Obtuse Margin 2, and Ramus Intermedius if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left Main coronary arteries. In order to accrue 109 subjects with significant Coronary Artery Disease as defined in the protocol, 826 subjects must be enrolled. Sample sizes provide 85% power with alpha of 0.05 for each statistical test.

ELIGIBILITY:
Subjects clinically indicated for nuclear stress test and who satisfy all the inclusion and exclusion criteria are eligible for participation.

Inclusion criteria:

Age 22 years or older Willing and able to give informed consent Clinical indication for nuclear stress test evaluation Chest pain syndrome

Two or more coronary artery disease risk factors as defined by:

1. Dyslipidemia: low-density lipoprotein (LDL) >130 mm/dL or high-density lipoprotein (HDL) <35 mm/dL or on treatment for dyslipidemia
2. Hypertension: blood pressure >140 millimeter of mercury (mmHg) systolic, >90 mmHg diastolic or on blood pressure altering treatment
3. Obesity: body mass index (BMI)>28
4. Current cigarette smoking
5. Diabetes: Type 1 or 2
6. Family history: coronary disease in a first or second degree relative

Exclusion criteria:

Body Mass Index (BMI)<18.5 or BMI >40

Known coronary disease as defined as:

Prior bypass surgery or coronary stenting Q-wave infarction on a past electrocardiogram (EKG) (>0.01 sec Q-wave duration in two adjacent leads)

Presence of pacemaker/defibrillator Presence of artificial valve Presence of obvious cyanotic or pre-diagnosed congenital heart defect and coarctation of the aorta Presence murmurs including valve lesions, ventricular septal defects, and arteriovenous (AV) fistulae.

Presence of moderate or severe valve disease as defined by >1/6 heart murmur on physical diagnosis Left Ventricular Assist Device (LVAD) Presence of scars on the site thorax areas Participation in trial within 30 days prior to collecting CADence data except participation in registry studies Asthma with wheezing Inability to lie flat in the supine position Acute coronary syndrome with elevated cardiac biomarkers (troponin (TP)>3x upper limit of normal (ULN) or creatine kinase MB (CKMB) >3x ULN) Heart Transplant Current cocaine use (within the past 24 hours, as reported by subject) Chronic Obstructive Pulmonary Disease (COPD) Contraindication to computed tomography (CT) angiography

* Renal failure with glomerular filtration rate (GFR)<50 (angio risk)
* Iodinated contrast allergy
* Elevated heart rate which cannot be controlled sufficiently to achieve a good computed tomography angiogram
* Body weight >350lbs.
* Sinus rhythm rate greater than 100 beats per minute at screening.
* Atrial fibrillation with average heart rate of greater than 70 beats per minute on resting screening electrocardiogram (ECG).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All enrolled subjects that received nuclear stress testing and either CT or standard coronary angiography after the CADence evaluation will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Thomas, MD, Study Chair — University of California, Los Angeles
Locations (24):
- United States (24):
  - University of Alabama, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Cardiology Associates of Mobile, Mobile, Alabama
  - UCLA, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular, Clearwater, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott/Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - HealthEast - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University, New York, New York
  - Mt. Sinai, New York, New York
  - North Ohio Research, Elyria, Ohio
  - Lancaster General, Lancaster, Pennsylvania
  - Jackson Clinic, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was held June 14, 2013 through February 10, 2016 at hospitals, clinics and research centers.
Groups:
- Overall Study: All patients enrolled in TURBULENCE study
Period: Overall Study
Arm/Group | Overall Study
Started | 1014
CADence Testing | 1013
Nuclear Stress Test | 992
CT and/or Standard Angiogram | 785
Completed | 785
Not Completed | 229
Not completed — Death | 1
Not completed — Lost to Follow-up | 66
Not completed — Physician Decision | 40
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 121

BASELINE CHARACTERISTICS:
Population: Baseline information was not provided for 3 of the 1,014 participants enrolled due to investigator withdrawals.
Arm/Group | Overall Study
Number analyzed (Participants) | 1011
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.14 (10.650)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486
  Male | 525
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 728
  Race/Ethnicity: Black or African American | 116
  Race/Ethnicity: Hispanic or Latino | 116
  Race/Ethnicity: Asian | 26
  Race/Ethnicity: Native American | 7
  Race/Ethnicity: Other | 18

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of CADence to Detect Stenosis Relative to SPECT Performance, Using Either CT or Standard Angiogram as the Gold Standard
Description: The CADence will be considered to have demonstrated effectiveness in detecting the presence of at least one lesion with ≥ 70% diameter stenosis anywhere in the proximal Left anterior Descending (pLAD), mid Left anterior Descending (mLAD), proximal Left Circumflex (pLCx), mid Left Circumflex (mLCx), proximal Right Coronary Artery (pRCA), mid Right Coronary Artery (mRCA), distal Right Coronary Artery (dRCA) and Obtuse Margin 1 (OM1), Obtuse Margin 2 (OM2), and Ramus Intermedius (RI) if segment diameter >2.5 mm or ≥50% diameter stenosis in the Left Main coronary arteries if sensitivity and specificity are non-inferior within 15 percentage points to a sensitivity of 83% and a specificity of 80%, which is the literature-based Objective Performance Criteria (OPC) for nuclear stress tests.
Time Frame: No more than 3 weeks between CADence, SPECT and standard or CT angiogram
Population: Per protocol subjects who completed all required testing and had analyzable results. Both Sensitivity and Specificity were assessed in this study.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Overall Study
Number analyzed (Participants) | 763
percent
  Sensitivity | 78 [76.1 to 90.8]
  Specificity | 36 [32 to 39]
Statistical Analysis 1: Comparison: Overall Study; The goal was to test the Sensitivity and specificity of CADence as compared to SPECT nuclear stress test OPC. Both were measured and reported in this study. The Sensitivity of CADence was 78% (95% CI 76.1-90.8%) while the specificity was 36% (95% CI 32-39%); Test type: Non-Inferiority — 15% equivalency margin against performance of SPECT nuclear stress test OPC. Both sensitivity and specificity were measured and the equivalency margin was set the same for both parameters.The goal was to test the Sensitivity and specificity of CADence as compared to SPECT nuclear stress test OPC. Both were measured and reported in this study. The Sensitivity of CADence was 78% (95% CI 76.1-90.8%) while the specificity was 36% (95% CI 32-39%); p = 0.012, Exact binomial test

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time CADence data was collected through completion of either their standard or computed tomography (CT) angiogram. The maximum time between CADence and either standard or CT angiogram was 6 weeks.
Description: An adverse event is considered serious if: 1) it results in death; 2) is life-threatening; 3) requires subject hospitalization or prolongation of existing hospitalization; 4) results in persistent or significant disability/incapacity; or 5) is an important medical event which may jeopardize the subject and may require medical or surgical intervention to prevent one of the previous outcomes.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 1/1014
Serious Adverse Events (participants affected / at risk) | 8/1014
Other Adverse Events (participants affected / at risk) | 10/1014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=1014)
Death (Congenital, familial and genetic disorders) | 1 (1) — Unknown cause of death, records unavailable. Died in sleep.
Unstable Angina (Cardiac disorders) | 1 (1)
Laryngoscopy (Surgical and medical procedures) | 1 (1) — History of vocal paralysis from stroke.
Knee Replacement (Surgical and medical procedures) | 1 (1) — Right total knee replacement
Pulmonary Embolism (Vascular disorders) | 1 (1)
Calcaneal Fractures (Injury, poisoning and procedural complications) | 1 (1) — Injury from a fall.
NSTEMI (Cardiac disorders) | 1 (1) — Non-ST-Elevation Myocardial Infarction (NSTEMI)
Epigastric Pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=1014)
CCTA-IV contrast infiltration (Surgical and medical procedures) | 5 (5) — Coronary Computed Tomography Angiography-Intravenous (CCTA-IV) contrast infiltration
CCTA-respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Wheezing/coughing after taking oral & iv metoprolol. Related to history of seasonal allergies and use of metoprolol.
CCTA-rash/hives (Skin and subcutaneous tissue disorders) | 2 (2) — Allergic reaction to contrast dye.
CCTA-symptomatic bradycardia (Cardiac disorders) | 1 (1)
Pleurisy (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days